CLINICAL TRIAL: NCT07112651
Title: The Effects of CL25216 on Vasomotor Symptoms in Women During Perimenopause: a Randomised, Double-blind, Placebo-controlled Study
Brief Title: Efficacy of CL25216 on Vasomotor Symptoms in Women During Perimenopause
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ApexCPG LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: APX/VMS/CL25216/25
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Vasomotor Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CL25216 (Experimental): 250 mg to take one capsule a day after breakfast for 105 days
  Interventions: Dietary Supplement: CL25216
- Placebo (Other): One capsule a day after breakfast for 105 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CL25216 — 250mg to take one capsule a day after breakfast for 105 days
  Arms: CL25216
Dietary Supplement: Placebo — One capsule a day after breakfast for 105 days
  Arms: Placebo

SUMMARY:
This study is to evaluate the effects of CL25216 on vasomotor symptoms in women during Perimenopause. Enrolled subjects will receive either CL25216 - 250 mg/day or placebo.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effects of CL25216 on vasomotor symptoms in women during perimenopause. A total of 80 female aged between40-55 years will be included in the study. Assessment of inclusion and exclusion criteria will be done based on clinical and laboratory investigations. The eligible subjects will be randomized as per the computer-generated randomization list. The subjects will be assigned to either CL25216 - 250 mg or placebo arms at 1:1ratio. The subjects will be instructed to take one capsule a day after breakfast for 105 days. Apart from primary and secondary outcomes, the study will also record the vital signs and adverse events to evaluate the herbal composition safety and tolerability. The safety assessment of the CL25216 will also include routine laboratory investigations on blood, urine and clinical chemistry at Screening/Randomisation visit and the final visit of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy overweight women (BMI: 25-29 kg/m2) aged between 40 to 55 years with reports of changes in their menstrual cycle for at least 3 months.
* Participants needed to have a total score of greater than 16 on the Greene Climacteric Scale (GCS), have an intact uterus and ovaries.
* Early Perimenopausal Women according "The Stages of Reproductive Aging Workshop (STRAW) Classification (-2)" irregular periods without skipping menstrual cycles and more than seven days difference in length of consecutive cycles.
* Subjects with serum FSH >20 U/L on 3-5 days of menstrual cycle.
* Subjects with normal pelvic TVS and breast mammogram.
* Subjects with normal fasting blood glucose level (<125 mg/dl).
* Subject understands the study procedures and provides signed informed consent to participate in the study.
* Subjects with normal blood thyroid profile.
* Females of childbearing potential who are sexually active must agree to use adequate contraception and can neither be pregnant nor lactating from screening throughout the duration of the study.
* Clinical screening including vital signs, electrocardiogram (ECG) and laboratory evaluations (including clinical chemistry, haematology, and complete urinalysis) within the reference range for the testing laboratory or the results are deemed not clinically significant for inclusion into this study by the investigator.

Exclusion Criteria:

* History of cerebrovascular disease, thrombo-embolic disorders, heart attack, or angina at any time or thrombophlebitis within the last 5 years, on anti-coagulant or anti-platelet drugs daily for any conditions.
* Subjects who had received hormonal treatment or any other herbal products in the previous 6 months.
* Subjects underwent treatment for COVID 19 within last 3 months or tested positive during the study will be excluded.
* Subjects diagnosed with ovarian cysts ≥ 4 cm or any underlying pathology in pelvic ultrasonography (USG) performed during screening.
* Chronic or acute life stressors relating to a major life change, experiencing depression and/or receiving medication for such illness or disorders, receiving statins or other drugs known to impact on steroid hormone levels.
* Subjects having active gall bladder disease, gynaecological or breast surgery in the last 6 months.
* History of breast, endometrial, other gynaecological cancer at any time or other cancer within the last 5 years.
* Subjects with abnormal ECG.
* Pregnant and breast feeding female.
* History of hypersensitivity reactions attributed to investigational product (IP) or its components or related products.
* Donation/loss of blood 1 unit or 350 mL within 90 days prior to receiving the first dose of study medication.
* Use of any recreational drugs (cocaine, amphetamine, barbiturates, benzodiazepines, cannabinoids, and morphine).
* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment, or compliance with the protocol.
* Participated in a clinical study with an investigational drug or biologic within the last 30 days.
* Any condition that in opinion of the investigator, does not justify the subjects" participation in the study.
* Subjects with a high blood pressure at screening (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥ 100 mmHg).
* Subjects with progressive systemic diseases (e.g. tuberculosis, leucosis, collagenosis, multiple sclerosis, AIDS, HIV infections, Hepatitis B surface antigen or Hepatitis C virus (HCV) antibodies or other auto-immune diseases).
* Evidence or history of clinically significant (in the judgment of the Investigator) haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neurologic diseases, or malignancies, hypothyroidism.
* High alcohol intake (>2 standard drinks per day), smokers (>5 cigarettes per day).

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy overweight women aged between 40 to 55 years
Enrollment: 80 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to the end of the study period in: Scores of Greene Climacteric Scale (GCS) | Day 1, 35, 70, and 105
  The Greene Scale is a validated instrument designed to provide a concise assessment of menopause symptoms. It consists of 21 items, each measuring the severity of climacteric symptoms on a scale from 0 (none) to 3 (severe), where 1 indicates mild and 2 indicates moderate symptoms. The total score ranges from 0 to 63, with higher scores reflecting more severe climacteric symptoms.

SECONDARY OUTCOMES:
Change from baseline to the end of the study period in: GCS sub-scale psychological symptoms | Day 1, 35, 70, and 105
  Psychological score is calculated from 1 to 11 items of GCS, ranges from 0 - 33, with higher scores reflecting more severe climacteric symptoms.
Change from baseline to the end of the study period in: GCS sub-scale scores: somatic/ physical symptoms | Day 1, 35, 70, and 105
  Somatic/ physical symptoms score is calculated from 12 to 18 items of GCS, ranges from 0 - 21, with higher scores reflecting more severe climacteric symptoms.
Change from baseline to the end of the study period in: GCS sub-scale scores: vasomotor symptoms. | Day 1, 35, 70, and 105
  Vasomotor symptoms score is calculated from 19 to 21 items of GCS, ranges from 0 - 9, with higher scores reflecting more severe climacteric symptoms.
Change from baseline to the end of the study period in: Resting Metabolic Rate (RMR) | Day 1, and 105
  RMR reflects the caloric expenditure necessary for life, without accounting for physical activity or digestion, measured by using metabolic analyzer. Increase in RMR is a sign of improved metabolism
Change from baseline to the end of the study period in: Positive and Negative Affect Schedule (PANAS-X) | Day 1, 35, 70, and 105
  The Positive and Negative Affect Schedule - Expanded Form (PANAS-X) is a validated self-report tool for assessing affective states, covering two broad dimensions: positive and negative affect. Each item has to be rated from 1 to 5 based on its severity. Each dimension is scored separately by summing the ratings of the individual items. As a result, the positive affect scale and the negative affect, with higher scores reflecting greater positive or negative affect, respectively.
Change from baseline to the end of the study period in: Quality of life questionnaire (Short Form -36) | Day 1, 35, 70, and 105
  The 36-Item Short Form (SF-36) is a self-reported questionnaire used to assess overall health and quality of life. It consists of 8 domains, each scored on a scale from 0 to 100. Higher scores indicate a better quality of life and improved health status.
Change from baseline to the end of the study period in: Sexual Function - Female Sexual Function Index (FSFI) | Day 1, 35, 70, and 105
  The FSFI was developed as a brief, easy-to-administer, self-report tool for assessing key dimensions or domains of sexual function and quality of life in various populations of women. Female Sexual Function Index (FSFI), a widely used tool with six domains (Arousal, Desire, Orgasm, Lubrication, Satisfaction, and Pain). The total FSFI score ranges from minimum score of 2 and maximum score of 36. Greater Scores indicates better sexual function
Change from baseline to the end of the study period in: The Hot Flush Weekly Weighted Score (HFWWS) | Day 1, 35, 70, and 105
  HFWW Score is calculated from a scale measuring the frequency and severity of hot flushes experienced daily for a week. Lower scores indicates better resolution of hot flushes
Change from baseline to the end of the study period in: Bodyweight | Day 1, 35, 70, and 105
  The subject's body weight is measured using a digital weighing scale. An improvement is indicated when the body weight falls within the normal range based on the subject's demographic characteristics.
Change from baseline to the end of the study period in: BMI | Day 1, 35, 70, and 105
  Body mass index is a calculated measure by considering the weight and height of a subject. A change in BMI from overweight to normal range is a positive indicator of healthy lifestyle.
Change from baseline to the end of the study period in: Scores of subjective self-assessments on hair quality | Day 1, 35, 70, and 105
  This is a subjective measurement of hair quality by considering the hair fall rate. The Highest Possible Score is 5.
Change from baseline to the end of the study period in: Skin wrinkle assessment | Day 1, 35, 70, and 105
  Visual assessment of skin wrinkles used to evaluate the appearance of skin aging and to determine the severity of wrinkles. This kind of assessment is typically done by a healthcare professional or dermatologist and involves examining the skin surface to identify and score wrinkles. Grade ranging from 0 to 9 where 0 represents no wrinkles and 9 represents deep wrinkles.
Change from baseline to the end of the study period in: Subject's self-assessment of skin Questionnaire | Day 1, 35, 70, and 105
  As the perception of the skin radiance is subjective, a self-assessment has been performed through a questionnaire. The scores range from 0 to 10, with higher scores indicating better skin quality in terms of complexion, smoothness, texture, elasticity, and hydration.
Change from baseline to the end of the study period in: Lipids | Day 1, and 105
  There is a clinically significant relationship between lipid metabolism and VMS like hot flashes and night sweats, especially in peri menopausal and postmenopausal women. Changes in lipid profiles may be both a cause and a consequence of hormonal shifts during this transition. Lower estrogen levels worsen lipid profiles and increases insulin resistance and central adiposity in perimenopusal/menopausal women.
Change from baseline to the end of the study period in: HOMA-IR | Day 1, and 105
  HOMA-IR is a simple and widely used method to estimate insulin resistance (IR) in perimenopause/menopause. HOMA-IR can be useful in assessing cardio metabolic risk in menopausal or postmenopausal women, especially those with vasomotor symptoms, which sometimes correlate with increased metabolic risk.
Change from baseline to the end of the study period in: FSH | Day 1, and 105
  It is a hormone produced by the pituitary gland and plays a crucial role in the reproductive systems of females. In perimenopause/menopause, the FSH level may rise disproportionately. Elevated FSH generally correlates with more frequent or severe hot flashes.
Change from baseline to the end of the study period in: LH | Day 1, and 105
  It is a hormone made by the pituitary gland that plays a key role in the reproductive system of females. In perimenopause/menopause, LH secretion becomes irregular and elevated, with occasional surges. Chronically elevated LH levels are seen in menopause.
Change from baseline to the end of the study period in: 17 beta-estradiol | Day 1, and 105
  17β-Estradiol (E2) is the most potent and biologically active form of estrogen in humans produced majorly by ovaries, followed by adrenal. Low estradiol is a key driver of VMS like hot flashes, night sweats, and sleep disturbances.
Change from baseline to the end of the study period in: AMH | Day 1, and 105
  AMH (Anti-Müllerian Hormone) is a marker of ovarian reserve, reflecting the number of remaining follicles in the ovaries. Levels decline with age and become undetectable at menopause. AMH testing could help identify women at risk for early and intense vasomotor symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Shree Hospitals, Vijayawada, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deecher DC, Dorries K. Understanding the pathophysiology of vasomotor symptoms (hot flushes and night sweats) that occur in perimenopause, menopause, and postmenopause life stages. Arch Womens Ment Health. 2007;10(6):247-57. doi: 10.1007/s00737-007-0209-5. Epub 2007 Dec 12. PMID 18074100
- [Background] Heger M, Ventskovskiy BM, Borzenko I, Kneis KC, Rettenberger R, Kaszkin-Bettag M, Heger PW. Efficacy and safety of a special extract of Rheum rhaponticum (ERr 731) in perimenopausal women with climacteric complaints: a 12-week randomized, double-blind, placebo-controlled trial. Menopause. 2006 Sep-Oct;13(5):744-59. doi: 10.1097/01.gme.0000240632.08182.e4. PMID 16894335
- [Background] Su HI, Freeman EW. Hormone changes associated with the menopausal transition. Minerva Ginecol. 2009 Dec;61(6):483-9. PMID 19942836
- [Background] Santoro N, Roeca C, Peters BA, Neal-Perry G. The Menopause Transition: Signs, Symptoms, and Management Options. J Clin Endocrinol Metab. 2021 Jan 1;106(1):1-15. doi: 10.1210/clinem/dgaa764. PMID 33095879
- [Background] Santoro N. Perimenopause: From Research to Practice. J Womens Health (Larchmt). 2016 Apr;25(4):332-9. doi: 10.1089/jwh.2015.5556. Epub 2015 Dec 10. PMID 26653408